CLINICAL TRIAL: NCT06560489
Title: Clinical Trial of Safety, Pharmacodynamics and Pharmacokinetic Characteristics of Multiple Subcutaneous Injections of LP-98 in Primary Treatment of HIV-infected Patients
Brief Title: Pharmacokinetics and Efficacy of Multiple Dosing of LP-98 for Injection in HIV-infected Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanxi Kangbao Biological Product Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KB_LP-98_102
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hiv
Keywords: LP-98; Double-Blind; Treatment-Naive HIV-Infected Individuals
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose level(1.25mg) (Experimental): This study consisted of 4 cohorts with 10 subjects in each group, who were randomly assigned to receive LP-98 treatment of 1.25 mg, 2.5 mg, 5 mg, and 10 mg. The method of administration was subcutaneous injection, and the interval of administration was 14 days, a total of 4 doses.
  Interventions: Drug: Subjects will be randomly assigned to receive 1.25 mg, 2.5 mg, 5 mg, or 10 mg of LP-98.
- Dose level(2.5mg) (Experimental): This study consisted of 4 cohorts with 10 subjects in each group, who were randomly assigned to receive LP-98 treatment of 1.25 mg, 2.5 mg, 5 mg, and 10 mg. The method of administration was subcutaneous injection, and the interval of administration was 14 days, a total of 4 doses.
  Interventions: Drug: Subjects will be randomly assigned to receive 1.25 mg, 2.5 mg, 5 mg, or 10 mg of LP-98.
- Dose level(5mg) (Experimental): This study consisted of 4 cohorts with 10 subjects in each group, who were randomly assigned to receive LP-98 treatment of 1.25 mg, 2.5 mg, 5 mg, and 10 mg. The method of administration was subcutaneous injection, and the interval of administration was 14 days, a total of 4 doses.
  Interventions: Drug: Subjects will be randomly assigned to receive 1.25 mg, 2.5 mg, 5 mg, or 10 mg of LP-98.
- Dose level(10mg) (Experimental): This study consisted of 4 cohorts with 10 subjects in each group, who were randomly assigned to receive LP-98 treatment of 1.25 mg, 2.5 mg, 5 mg, and 10 mg. The method of administration was subcutaneous injection, and the interval of administration was 14 days, a total of 4 doses.
  Interventions: Drug: Subjects will be randomly assigned to receive 1.25 mg, 2.5 mg, 5 mg, or 10 mg of LP-98.

INTERVENTIONS:
Drug: Subjects will be randomly assigned to receive 1.25 mg, 2.5 mg, 5 mg, or 10 mg of LP-98. — This study consisted of 4 cohorts with 10 subjects in each group, who were randomly assigned to receive LP-98 treatment of 1.25 mg, 2.5 mg, 5 mg, and 10 mg. The method of administration was subcutaneous injection, and the interval of administration was 14 days, a total of 4 doses.

SUMMARY:
A Randomized, Double-Blind, Parallel-Group, Exploratory Clinical Study to Evaluate the Safety, Pharmacodynamic Effects, and Pharmacokinetic Characteristics of Multiple Subcutaneous Injections of LP-98 in Treatment-Naive HIV-Infected Individuals

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallelize-designed, multicenter, exploratory clinical study to evaluate the safety, PD, and PK profile of multiple subcutaneous injections of LP-98 in HIV-infected individuals who have not received antiviral therapy.

This study consisted of 4 cohorts with 10 subjects in each group, who were randomly assigned to receive LP-98 treatment of 1.25 mg, 2.5 mg, 5 mg, and 10 mg. The method of administration was subcutaneous injection, and the interval of administration was 14 days, a total of 4 doses.

The study included screening period (D-28~D-1), treatment period (D1-D57), and follow-up period (D58~D71).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and obtain informed consent prior to any study-related evaluation;
2. Aged 18-65 years at the time of the screening visit (including the cut-off), male or female;
3. At the time of screening visit, the weight of male subjects is not less than 50 kg and that of female subjects is not less than 45 kg;
4. Plasma HIV RNA level ≥1000 copies /mL, CD4+T lymphocyte count ≥200 /μL;
5. For female subjects: Only subjects with no reproductive potential were included, including surgical sterilization at least 6 weeks prior to the screening visit (documented hysterectomy or bilateral oopectomies), and menopause ≥12 months prior to the screening visit (menopause confirmed by follicle stimulating hormone (FSH) level ≥40IU/L);
6. For male subjects with fertile female partners, consent must be given to the use of non-drug contraception for 14 days prior to dosing, during the study period, and for 3 months after dosing. Male subjects are not allowed to donate sperm during this period;
7. Be willing to comply with visits, study treatments, laboratory tests, and other study-related procedures and requirements as specified in the study protocol.

Exclusion Criteria:

1. is allergic to the investigational drug product or its excipients, or has a history of severe allergy (including any food allergy or drug allergy);
2. have received antiviral therapy (ART), or been vaccinated against HIV;
3. Have a history of serious illness or other serious chronic diseases;
4. Have a history of mental illness, or have a family history of mental illness;
5. any of the following conditions exist: i. Unexplained persistent irregular fever above 38 °C within 1 month before or during the screening period; ii. Persistent diarrhea (more than 3 stools/day) within 1 month before or during the screening period; iii. Severe infection, opportunistic infection, or sepsis in the 6 months prior to or during the screening period;
6. Hepatitis B surface antigen (HBsAg) positive, or hepatitis C antibody (HCV-Ab) positive;
7. The 12-lead ECG was abnormal and clinically significant during screening, such as QTcF interval (Fridericia correction) > 450 ms in male and > 470 ms in female;
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 1.5 times ULN, or total bilirubin > 1.5 times ULN during screening;
9. Serum creatinine clearance (Ccr) at screening was < 60 mL/min (calculated according to Cockcroft-Gault formula);
10. A known or suspected history of drug abuse (morphine, methamphetamine, ketamine, dimethylene dioxyamphetamine, THC, cocaine), or a positive baseline drug screening test;
11. Heavy drinking in the year before screening (drinking more than 14 standard units per week, 1 standard unit containing 14 g of alcohol, such as 5% beer 360 ml, 40% spirits 45 ml, 12% wine 120 ml); Or fail to comply with the no-alcohol policy for the duration of the study;
12. Smoking more than 5 cigarettes per day in the 3 months prior to screening, or failing to comply with the no-smoking policy during the study period;
13. have received any vaccine in the three months prior to screening, or plan to receive any vaccine during the study period;
14. received any investigational drug therapy or participated in any drug/investigational device trial within 3 months prior to dosing;
15. had undergone a major surgical procedure within 30 days prior to dosing or planned to undergo a major surgical procedure during the study period;
16. Those who have donated blood or lost blood ≥ 400 ml or received blood transfusion within 3 months before screening;
17. There are other circumstances that are not suitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in respiration rate of Vital Signs. | Within 71 days after the first administration.
  Respiration rate in times / minute
Changes from baseline in blood pressure of Vital Signs. | Within 71 days after the first administration.
  Blood pressure in mmHg
Changes from baseline in Blood lactate of Laboratory Examination. | Within 71 days after the first administration.
  Changes of blood lactate will be recorded.
Changes from baseline in body temperature of Vital Signs. | Within 71 days after the first administration.
  Body temperature in Celsius degree
Changes from baseline in red blood cell count of Laboratory Examination. | Within 71 days after the first administration.
  Red blood cell count in whole blood is reported in the form of number.
Changes from baseline in white blood cell count of Laboratory Examination. | Within 71 days after the first administration.
  White blood cell count in whole blood is reported in the form of number.
Changes from baseline in neutrophil count of Laboratory Examination. | Within 71 days after the first administration.
  Neutrophil count in whole blood is reported in the form of number.
Changes from baseline in lymphocyte count of Laboratory Examination. | Within 71 days after the first administration.
  Lymphocyte count in whole blood is reported in the form of number.
Changes from baseline in platelet count of Laboratory Examination. | Within 71 days after the first administration.
  Platelet count in whole blood is reported in the form of number.
Changes from baseline in hemoglobin of Laboratory Examination. | Within 71 days after the first administration.
  Changes of hemoglobin concentration（g/dL）in whole blood will be recorded.
Changes from baseline in PT of Laboratory Examination. | Within 71 days after the first administration.
  Prothrombin time (PT) is a screening test for exogenous coagulation factors.
Changes from baseline in INR of Laboratory Examination. | Within 71 days after the first administration.
  International standardized ratio (INR) is calculated from prothrombin time and international sensitivity index (ISI) of the reagent.
Changes from baseline in APTT of Laboratory Examination. | Within 71 days after the first administration.
  Activated partial thromboplastin time (APTT) is a screening test for endogenous coagulation factors.
Changes from baseline in total bilirubin of Laboratory Examination. | Within 71 days after the first administration.
  Changes of total bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in direct bilirubin of Laboratory Examination. | Within 71 days after the first administration.
  Changes of direct bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in ALT of Laboratory Examination. | Within 71 days after the first administration.
  Changes of ALT concentration (U/L) in serum will be recorded.
Changes from baseline in AST of Laboratory Examination. | Within 71 days after the first administration.
  Changes of AST concentration (U/L) in serum will be recorded.
Changes from baseline in total protein of Laboratory Examination. | Within 71 days after the first administration.
  Changes of total protein concentration (g/L) in serum will be recorded.
Changes from baseline in albumin of Laboratory Examination. | Within 71 days after the first administration.
  Changes of albumin concentration (g/L) in serum will be recorded.
Changes from baseline in urea of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urea concentration (mmol/L) in serum will be recorded.
Changes from baseline in creatinine of Laboratory Examination. | Within 71 days after the first administration.
  Changes of creatinine concentration (μmol/L) in serum will be recorded.
Changes from baseline in uric acid of Laboratory Examination. | Within 71 days after the first administration.
  Changes of uric acid concentration (μmol/L) in serum will be recorded.
Changes from baseline in glucose of Laboratory Examination | Within 71 days after the first administration.
  Changes of glucose concentration (mmol/L) in serum will be recorded.
Changes from baseline in potassium of Laboratory Examination. | Within 71 days after the first administration.
  Changes of potassium concentration (mmol/L) in serum will be recorded.
Changes from baseline in sodium of Laboratory Examination. | Within 71 days after the first administration.
  Changes of sodium concentration (mmol/L) in serum will be recorded.
Changes from baseline in chlorine of Laboratory Examination. | Within 71 days after the first administration.
  Changes of chlorine concentration (mmol/L) in serum will be recorded.
Changes from baseline in urine specific gravity of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urine specific gravity will be recorded.
Changes from baseline in urine pH of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urine pH value will be recorded.
Changes from baseline in urine glucose of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urine glucose will be examined by qualitative test (positive or negative).
Changes from baseline in urine protein of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urine protein will be examined by qualitative test (positive or negative).
Changes from baseline in urine ketone body of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urine ketone body will be examined by qualitative test (positive or negative).
Changes from baseline in urine white blood cell of Laboratory Examination. | Within 71 days after the first administration.
  Changes of white blood cell in urine will be examined by qualitative test (positive or negative).
Changes from baseline in urine bilirubin of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urine bilirubin will be examined by qualitative test (positive or negative).
Changes from baseline in urine occult blood of Laboratory Examination. | Within 71 days after the first administration.
  Changes of urine occult blood will be examined by qualitative test (positive or negative).
Changes from baseline in Electrocardiogram. | Within 71 days after the first administration.
  The cardiac rhythm is showed in electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded，To evaluate the incidence of abnormal electrocardiogram.
Changes from baseline in CK of Laboratory Examination | Within 71 days after the first administration.
  Changes of CK concentration (U/L) in serum will be recorded.
Changes from baseline in CK-MB of Laboratory Examination | Within 71 days after the first administration.
  Changes of CK-MB concentration (ng/mL) in serum will be recorded.
Changes from baseline in LDH of Laboratory Examination | Within 71 days after the first administration.
  Changes of LDH concentration (U/L) in serum will be recorded.
Changes from baseline in ALP of Laboratory Examination | Within 71 days after the first administration.
  Changes of ALP concentration (U/L) in serum will be recorded.
Changes from baseline in Triglyceride of Laboratory Examination | Within 71 days after the first administration.
  Changes of Triglyceride concentration (mmol/L) in serum will be recorded.
Changes from baseline in CHOL of Laboratory Examination | Within 71 days after the first administration.
  Changes of CHOL concentration (mmol/L) in serum will be recorded.
Changes from baseline in TP of Laboratory Examination | Within 71 days after the first administration.
  Changes of TP concentration (g/L) in serum will be recorded.
Changes from baseline in ALB of Laboratory Examination | Within 71 days after the first administration.
  Changes of ALB concentration (g/L) in serum will be recorded.
Changes from baseline in UA of Laboratory Examination | Within 71 days after the first administration.
  Changes of UA concentration (μmol/L) in serum will be recorded.

SECONDARY OUTCOMES:
Changes from baseline in Immunogenic blood collection of Laboratory Examination. | Within 71 days after the first administration.
  Changes of immunogenic blood collection will be recorded.The historical changes of test results (including positive rate and titer) of various indicators were counted.
Changes from baseline in HIV viral load detection of Laboratory Examination. | Within 71 days after the first administration.
  Changes of HIV viral load detection will be recorded.
Changes from baseline in CD4+T cell counts of Laboratory Examination. | Within 71 days after the first administration.
  Changes of CD4+T cell counts will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Qingxia Zhao, Doctor, Study Director — Henan Provincial Hospital for Infectious Diseases (Zhengzhou Sixth People's Hospital)
Locations (1):
- Henan Provincial Hospital for Infectious Diseases (Zhengzhou Sixth People's Hospital), Zhengzhou, Henan, China